CLINICAL TRIAL: NCT01564420
Title: Pharmacokinetic/Pharmacodynamic Modeling of Morphine for Postoperative Analgesia Through a Patient Controlled Device After Coronary Artery Bypass Grafting. Intrathecal Morphine Significantly Reduces Drug Consumption
Brief Title: Morphine Postoperative Analgesia and Pharmacokinetic/Pharmacodynamic Modeling
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Silvia Regina Cavani Jorge Santos, Chair Professor, University of Sao Paulo
Other Study IDs: Santos 2012
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Cardiopulmonar Artery Bypass Grafting
Keywords: pharmacokinetic/pharmacodynamic modeling; intrathecal morphine; postoperative analgesia; patient-controlled analgesia device

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For pharmacokinetic analysis, a serial of blood samples of patients was collected postoperatively after the extubation from a venous catheter (5mL each) into an EDTA tube (BD, Sao Paulo/Brazil) in the periods as follows: 0, 0.08, 0.25, 0.5, 1, 3, 6, 12, 18, 24 and 36 hrs. Blood samples were centrifuged at 2800 g for 20 minutes, plasma was transferred to labeled polyethylene vials and frozen at -80ºC until drug plasma assay.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intrathecal morphine: Patients were randomized for general anesthesia, and allocated in the control group and morphine intrathecal group.
- Control group

SUMMARY:
The currently available data are insufficient to develop a model that achieves optimum morphine dose individualization at the postoperative period of coronary artery bypass grafting (CABG). Therefore, the objective of the study was to apply a PK/PD model that could justify morphine consumption, drug plasma concentration and pain intensity during the postoperative period after CABG and evaluate the post operative pain.

DETAILED DESCRIPTION:
The protocol was a prospective, open-label study, approved by the institutional ethical committee of the hospital where the study was performed. Patients were randomly assigned to receive general anesthesia plus intrathecal morphine at a dosage of 400 mcg (morphine group) or general anesthesia alone (control group) according to a simple computer-generated list.

ELIGIBILITY:
Inclusion Criteria:

* eligible to cardiopulmonary artery bypass grafting surgery

Exclusion Criteria:

* fraction of ejection below 40%
* contraindications to neuraxial blockage
* coagulopathy
* use of low-weight heparin
* warfarin or a platelet aggregation inhibitor other than aspirin,
* systemic or local infection
* and patients with a specific contraindication on the medication employed in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease, eligible to cardiopulmonary artery bypass grafting surgery
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2003-01; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | two days
  From the end of surgery until 36 hours of postoperative period
PK/PD modelling | 2 days
  From the begin of surgery until 36 hours of postoperative period

SECONDARY OUTCOMES:
PK parameter: Cmax (peak plasma concentration) | 2 days
  from the begin of surgery until 36 hours of postoperative period
PK parameter: Tmax (time to achieve the maximum concentration) | 2 days
  from the begin of surgery until 36 hours of postoperative period
PK parameter: AUC (area under the plasma cocentration versus time curve) | 2 days
  from the begin of surgery until 36 hours of postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Silvia RCJ Santos, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Pharmaceutical Science, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] dos Santos LM, Santos VC, Santos SR, Malbouisson LM, Carmona MJ. Intrathecal morphine plus general anesthesia in cardiac surgery: effects on pulmonary function, postoperative analgesia, and plasma morphine concentration. Clinics (Sao Paulo). 2009;64(4):279-85. doi: 10.1590/s1807-59322009000400003. PMID 19488583
- See also: Group web site — http://www.anestesiologiausp.com.br
- See also: Health national council web site — http://conselho.saude.gov.br/web_comissoes/conep/index.html